CLINICAL TRIAL: NCT01106365
Title: Repetitive Deep Transcranial Magnetic Stimulation in Multiple Sclerosis - A Pilot Study to Evaluate Safety and Efficacy of Deep rTMS on Fatigue and Depressivity in Patients With Multiple Sclerosis
Brief Title: Repetitive Deep Transcranial Magnetic Stimulation in Multiple Sclerosis
Acronym: rTMS in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Friedemann Paul, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rTMS in MS
Record Dates: First submitted 2010-04-16; First posted 2010-04-19 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; fatigue; depressivity; repetitive deep transcranial magnetic stimulation
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- prefrontal cortex (PFC) (Experimental): rTMS with the H-coil to the prefrontal cortex (PFC)
  Interventions: Device: H-coil (Repetitive deep transcranial magnetic stimulation)
- motor cortex (Active Comparator): rTMS with the H-coil to the motor cortex
  Interventions: Device: H-coil (Repetitive deep transcranial magnetic stimulation)
- sham treatment (Sham Comparator): sham treatment
  Interventions: Device: H-coil (Repetitive deep transcranial magnetic stimulation)

INTERVENTIONS:
Device: H-coil (Repetitive deep transcranial magnetic stimulation) — Repetitive deep transcranial magnetic stimulation of prefrontal cortex or motor cortex or sham stimulation
  Other Names: H-coil (Brainsway LTD., 19 Hartom Str., Jerusalem, Israel)

SUMMARY:
Multiple sclerosis (MS) is a chronic-inflammatory autoimmune central nervous system disorder and a leading cause of neurological disability in younger adults in Western countries. Besides "classic" neurological symptoms both depressivity and fatigue are among the most frequent symptoms in MS, affecting up to 90% of patients at onset or during the course of the disease. Neither are the psychological and immunological backgrounds of both well understood, nor are there numerous controlled therapeutic trials which would offer convincing treatment options for fatigue and depressivity in MS.

Transcranial magnetic stimulation (TMS) has been frequently used to investigate altered hemispheric and inter-hemispheric connectivity in MS. Recently, first therapeutic trials have been performed to address specific MS-related symptoms by TMS. Koch et al. demonstrated an improvement of hand dexterity following repetitive TMS, and Centonze and colleagues showed reduced spasticity following TMS.

Recently, a specific coil for the stimulation of deeper brain regions including the deep nuclei was developed, the so-called H-coil. It successfully stimulates deeper (pre-frontal) brain regions. Stimulation with this coil has been shown to be safe and well tolerated in healthy volunteers, and in patients suffering from major depression.

The aim of this project is to apply deep TMS with the H-coil to the prefrontal cortex (PFC) of MS patients. The PFC is the region at which stimulation is aimed in previous depression studies as this brain region has been shown to play a relevant role in affective disorders. It is the primary aim of this study, to evaluate the safety and tolerability of deep TMS with the H-coil in MS patients with fatigue or depressivity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with clinically definite MS according to Polman
* Age 18 to 60
* EDSS 0 to 6
* Relapse-free > 30 days prior to inclusion
* Stable immunomodulatory or immunosuppressive therapy or treatment-naïve for > 3 months prior to inclusion
* In case of treatment with antidepressants: stable therapy > 3 months
* A score of ≥ 4 on the FSS (fatigue severity scale)8 or
* A score of ≥ 12 on the Beck Depression Inventory (BDI)
* Highly effective methods of birth control for females

Exclusion Criteria:

* Personal or family history of epilepsy, brain tumor, brain injury
* History of metallic particles in the eye or head outside the mouth
* Cardiac pacemakers, implanted neurostimulators, cochlear implants, implanted medication pumps
* History of drug or alcohol abuse
* Pregnancy
* Relapse of MS < 30 days prior to inclusion
* I.v. corticosteroid treatment < 30 days prior to inclusion
* Change of immunomodulatory therapy < 30 days prior to inclusion
* Change of antidepressant therapy < 3 months prior to inclusion
* Comedication with neuroleptics and tricyclic antidepressants (amitriptyline etc.) during the entire study
* patients with increased intracranial pressure (which lowers seizure threshold)
* intracardiac lines
* significant heart disease
* bipolar disorder
* history of stroke or other brain lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety | 3x/week during treatment phase
  examination by physician, assessement of adverse events

SECONDARY OUTCOMES:
Fatigue | 3x/week during treatment period
  Assessment of Fatigue via Fatigue Severity Scale FSS
Depressivity | 3x/week during treatment period
  Assessment of Depressivity via Beck Depression Inventory BDI

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University Berlin (NeuroCure Clinical Research Center NCRC), Berlin, Germany

REFERENCES:
- [Result] Gaede G, Tiede M, Lorenz I, Brandt AU, Pfueller C, Dorr J, Bellmann-Strobl J, Piper SK, Roth Y, Zangen A, Schippling S, Paul F. Safety and preliminary efficacy of deep transcranial magnetic stimulation in MS-related fatigue. Neurol Neuroimmunol Neuroinflamm. 2017 Dec 13;5(1):e423. doi: 10.1212/NXI.0000000000000423. eCollection 2018 Jan. PMID 29259998